CLINICAL TRIAL: NCT03491982
Title: Compliance Feasibility Study for Remote Phase 2 Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Lisa Alderson MD, F.A.C.C., Assistant Professor, St. Louis University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 28544
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Referred by Cardiologist for Phase 2 Cardiac Rehabilitation
Keywords: Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Remote Cardiac Rehab — Remote Cardiac Rehab

SUMMARY:
This study evaluates the compliance of patients in a Phase 2 (outpatient clinic based) cardiac rehabilitation program, who are offered the opportunity to perform the rehab remotely (e.g. at home, not at the clinic), using a remote monitor and smart-phone application.

DETAILED DESCRIPTION:
In spite of the fact that cardiac rehabilitation has been shown to be beneficial to patients who have had a cardiac event, such as a heart attack, only 5% of eligible patients complete this program. Some of the reasons cited include limited facility access, travel time and cost.

We are testing the hypothesis that cardiac rehab compliance will be greater if patients are offered the opportunity, and associated technology, to perform cardiac rehab anywhere.

ELIGIBILITY:
Inclusion Criteria:

* referred to SLU cardiac rehab facility

Exclusion Criteria:

* does not own app compatible smart phone
* dementia
* syncope
* valvular disease
* life expectancy < 1 year
* non-English speaking
* unstable angina
* decompensated congestive heart failure
* ventricular arrhythmia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients completing remote rehab program compared to case controls | Immediately after cardiac rehab completion or stoppage

SECONDARY OUTCOMES:
Six minute walk test compared to case controls | Immediately after cardiac rehab completion or stoppage
depression score vs case controls | Immediately after cardiac rehab completion or stoppage
Average number of minutes in exercise rehab compared to case controls | Immediately after cardiac rehab completion or stoppage

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Alderson, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University - SLUCare, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
no current plan